CLINICAL TRIAL: NCT03879382
Title: A Phase I Clinical Trial of Human CD19/BCMA Bispecific CAR-T Cell Therapy for Subjects With Relapsed and Refractory POMES Syndrome.
Brief Title: Anti-CD19/BCMA Bispecific CAR-T Cell Therapy for R/R POMES
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRain-POMES01
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: POMES Syndrome; Relapsed and Refractory POMES Syndrome
Keywords: CD19/BCMA; Bispecific CAR-T Cell; POMES Syndrome; Relapsed and Refractory
MeSH Terms: conditions — Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/BCMA CAR-T cells (Experimental): Administration with anti-CD19/BCMA CAR-T cells in the relapsed and refractory POMES Syndrome patients
  Interventions: Biological: anti-CD19/BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: anti-CD19/BCMA CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-CD19 and anti-BCMA CARs
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 300mg/m2/d

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-CD19/BCMA bispecific chimeric antigen receptors (CARs) T cell therapy for relapsed and refractory POMES Syndrome.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the feasibility ad safety of anti-CD19/BCMA CAR-T cells in treating patients with relapsed and refractory POMES Syndrome.

Secondary Objectives

1. To access the efficacy of anti-CD19/BCMA CAR-T cells in patients with POMES Syndrome.
2. To determine in vivo dynamics and persistency of anti-CD19/BCMA CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival > 12 weeks;
* Diagnosis of POMES Syndrome;
* The criteria for relapsed and refractory POMES Syndrome: patients previously received at least 3 different prior treatment regimens for multiple myeloma, including Alkylating agent and other protein inhibitors (eg: Bortezomib), and have disease progression in the past 60 days;
* At least 90 days after stem cell transplantation;
* Creatinine≤2.0 mg/dl;
* Bilirubin≤2.0 mg/dl;
* The ALT/AST value is lower than 2.5-fold of normal value;
* Accessible to intravenous injection, and no white blood cell collection contraindications;
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 30 days after the CTL infusion. Male partner should use a condom;
* 5mg/day dose of Prednisone or other equivalent steroid hormone drugs (eg: Dexamethasone) were not used for two weeks before apheresis and CAR-T infusion;
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

* • In the first 5 years before screening, there are malignant tumors other than POMES Syndrome, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery，and catheter carcinoma in situ after radical surgery;

  * Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA titer higher than the upper limit of detection; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency Viral (HIV) antibody positive; Positive syphilis test;
  * Any unstable systemic disease including, but not limited to, active infection (except for local infection), unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmia, liver, kidney or metabolic disease requiring medication;
  * Any other diseases could affect the outcome of this trial;
  * Any affairs could affect the safety of the subjects or outcome of this trial;
  * Pregnant or lactating women, or planned pregnancy during treatment or within 1 year after treatment, or a male subject whose partner plans pregnancy within 1 year of their cell transfusion;
  * Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
  * Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
  * Received CAR-T treatment or other gene therapies before enrollment;
  * Patients with symptoms of central nervous system or brain metastasis or have received treatment for central nervous system or brain metastasis (radiotherapy, surgery or other treatment) within 3 months before enrollment;
  * Subject suffering disease affects the understanding of informed consent or comply with study protocol;
  * The investigators consider other conditions unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 6 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for POMES Syndrome | 8 weeks
  Overall complete remission rate defined by the standard response criteria for POMES Syndrome
Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No